CLINICAL TRIAL: NCT04234763
Title: Metabolomics Determinant of Postprandial Metabolism Following Meal-Challenge Test in Diabetes State Using NMR-based Metabolomics Approach
Brief Title: Postprandial Metabolites of Meal Challenge Test in Diabetes State
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Barakatun Nisak Bt Mohd Yusof, Associate Professor, Universiti Putra Malaysia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 9613400
Record Dates: First submitted 2019-12-03; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Type2 Diabetes; Postprandial Hyperglycemia
Keywords: Glycemic Index; NMR metabolomics; Postmeal glucose
MeSH Terms: conditions — Hyperglycemia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The meal challenge test (MCT) models are designed to be high glycemic index (GI) (GI=63, GL=25) and low GI meal (GI=46, GL=16), isocaloric (300kcal) with identical macronutrient distribution. The meals will be prepared on the morning of the test, portioned by weighing and served warm.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T2D patients (Experimental): T2D patients (n=24) will be randomized to high GI and low GI MCT randomly.
  Interventions: Behavioral: Strategies to lower postprandial hyperglycemia in T2D patients
- Healthy individuals (Active Comparator): Healthy individuals (n=24) will be randomized to high GI MCT only.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Strategies to lower postprandial hyperglycemia in T2D patients — T2D patients will undergo a 14-day chronic feeding trial intervention where the strategies to lower postprandial hyperglycemia will be educated. For example, to control portion of carbohydrate, incorporate low GI food and diabetes-specific formula, promote physical activity and practice consistent meal timing. After that, patients will undergo MCT again to evaluate the difference before and after the intervention.
  Arms: T2D patients
Behavioral: Control group — Assess nutritional status and no active intervention is conducted.
  Arms: Healthy individuals

SUMMARY:
Postprandial hyperglycemia is a hallmark feature of Type 2 Diabetes Mellitus (T2D), and persistent elevated glycemic level has shown to be strongly associated with oxidative stress, and a risk factor for cardiovascular disease (CVD). In Malaysia, the glycemic control is poor and patients with T2D commonly experiencing persistent postprandial hyperglycemia (12.7 mmol/L). A low glycemic index (GI) meal has been reported to reduce postprandial glycemia and insulin concentration in patients with T2D. Metabolomics technique can be used to identify comprehensive metabolites in response to different diet. Till date, local scientific data documented on the role and interaction between diet and metabolites for the Malaysian patients with T2D is unknown. This study is to determine the postprandial metabolomic effect of low and high GI meals in patients with T2D using the NMR-based metabolomics approach. Then, patients with T2D will be assigned for 14 days of chronic feeding trial intervention. This study will help to establish local baseline data and understand the impact of meal-patterns on metabolic and metabolite at postprandial responses.

DETAILED DESCRIPTION:
Despite targeting to optimize fasting blood glucose and lowering HbA1c level, postprandial hyperglycemia needs to be highlighted in the management of Type 2 Diabetes Mellitus (T2D). Postprandial hyperglycemia is the rapid and significant rise in blood glucose level above 7.8 mmol/L 2 hour after meal ingestion. It is strongly associated with oxidative stress and a risk factor for cardiovascular disease (CVD).

In Malaysia, the glycemic control is poor, and patients with T2D commonly experiencing persistent hyperglycemia (12.7 mmol/L), which is the highest concentration in South East Asia region. Nonetheless, a low glycemic index (GI) meal has been reported to reduce postprandial glycemia and insulin concentration in patients with T2D but the metabolite responsiveness following low GI meal is not studied yet. The study of the postprandial state is imperative as it reveals multiple aspects of metabolic health that would not be apparent from solely studying the fasting parameters.

Hence, the objective of this study is to determine the postprandial metabolomic effects of low and high GI meals in patients with T2D using the NMR-based metabolomics approach. Then, the postprandial metabolic response and metabolomic profiles before and after the 14 days chronic feeding trial intervention will be determined and compared. The calculated sample size was 24 patients with T2D and 24 healthy individuals. The study design for meal challenge test (MCT) is a single-blinded, randomized crossover trial with 1-week washout period; whereas a case-control design will be used to compare metabolomic profiles of patients with T2D and healthy individuals.

The MCT model is designed to be high GI (63) and low GI (46) with similar caloric value. During the test day, participants are required to consume the meal within 15 minutes and the blood sample will be taken at the following time points: 0min (fasting), 30, 60, 120, 180 and 240 min. Meanwhile, the urine sample will also be collected at 0, 60 and 240 min accordingly.

The blood sample will be analyzed for blood glucose, insulin, GLP-1, and metabolites; while the urine sample will be analyzed for metabolites. The findings of this study are able to provide fundamental data on metabolic responsiveness of T2D patients following specific meal-plan tailored to Malaysian meal pattern using NMR-based metabolomics approach. Besides, this study is able to establish a local baseline data of postprandial metabolite profiles of patients with T2D following a specific meal plan. At the same time, this study contributes insight to improve diabetes meal-plan that is friendly to postprandial metabolic perturbations.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-35.0 kg/m²
* Glycemic control (HbA1c level 6.5 - 10.0%)
* On stabilised oral-antidiabetic drug (OAD) : metformin, sulphonylureas, SGLT2 inhibitors
* Estimated glomerular filtration rate (GFR) >60ml/min
* No clinically significant cardiovascular, renal or liver disease

Exclusion Criteria:

* Smokers
* Pregnant and lactating women
* Food allergies or intolerances
* On weight loss diet
* On insulin therapy
* On OAD: DPP-4 inhibitors, GLP-1 receptor agonists, acarbose
* Anemia (Hb <10g/dL)
* On regular use of hormones or anti-inflammatory medication (aspirin, corticosteroid)
* Suggestive indicators for impaired thyroid (high T2H level) or liver function

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Postprandial glucose | Change from baseline and after 14-days intervention
  Between low GI and high GI meal challenge measured by blood plasma using Abbott Architect c16000 analyser
Postprandial insulin | Change from baseline and after 14-days intervention
  Between low GI and high GI meal challenge measured by blood serum using COBAS e411 analyzer
Postprandial GLP-1 | Change from baseline and after 14-days intervention
  Between low GI and high GI meal challenge measured by blood plasma using total ELISA kit
1H-NMR metabolites | Change from baseline and after 14-days intervention
  Between low GI and high GI meal challenge measured by blood plasma using 1H-NMR spectrometer
Postprandial 1H-NMR metabolites | During the 4 hour meal challenge
  Between T2D and healthy individuals measured by blood plasma using 1H-NMR spectrometer

SECONDARY OUTCOMES:
Body mass index (BMI) | Before and after the 14-days intervention
  Measured by weight change using Tanita digital weighing scale
Waist circumference | Before and after the 14-days intervention
  Using measuring tape
Lipid profile | Before and after the 14-days intervention
  Measured by blood plasma using Abbott Architect c16000 analyser
Dietary glycemic index (GI) | Before and after the 14-days intervention
  Between T2D and healthy individuals measured using Dietary History Questionnaire
Dietary Glycemic load(GL) | Before and after the 14-days intervention
  Between T2D and healthy individuals measured using Dietary History Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Assoc. Prof. Dr. Barakatun Nisak, Principal Investigator — Faculty of Medicine and Health Sciences, Universiti Putra Malaysia
Locations (1):
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No